CLINICAL TRIAL: NCT02566954
Title: 3 Dimensional Study of Lower Limbs and Feet of Children in Standing Position
Acronym: MI3DEOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Lenval (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 14-HPNCL-03
Record Dates: First submitted 2015-07-22; First posted 2015-10-02 (Estimated); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: Limb Deformities
Keywords: radiology; 3D measurement; lower limb

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 3D measurement of the lower limb by EOS (Experimental): The intervention is to performed an additional radiologic exam by the EOS® system of imaging. This imaging is not usually realized for the patient.
  3 dimensional study of lower limbs and feet of children in standing position will be performed using the EOS® system (EOS® Imaging, France)
  Interventions: Other: 3D measurement of the lower limb by EOS

INTERVENTIONS:
Other: 3D measurement of the lower limb by EOS — The intervention is to performed an additional radiologic exam by the EOS® system of imaging. This imaging is not usually realized for the patient.
  3 dimensional study of lower limbs and feet of children in standing position will be performed using the EOS® system (EOS® Imaging, France)

SUMMARY:
The study will be in 3 parts: first one will be to address the key question of the lower limb frontal alignment based on both three-dimensional measurements of low-dose bi-planar X-rays and foot morphology assessment. Indeed, a major issue in the management of lower limb disorders is the ability to correctly assess abnormal development and decide on the most adapted treatment option. In particular, the link between lower limb disorders and foot morphology remain unclear. Recently, quantitative 3D measurement of the lower limb in children has been successfully assessed using low-dose biplanar X-rays.

Second part will be to assess the reproducibility of the 3dimensional reconstructions whether they are made by a radiology technician, or by a so-called expert through collecting datas from 3 centers of pediatric surgery where EOS Imaging system is daily used to get spine or lower limb X-Rays.

Last part will be to work on the recently developed weight-bearing foot 3D reconstruction method for clinical use using the Parametric Personalized Modelling approach (PPM). This will allow having a better understanding and evaluation of foot's anatomy and patho-anatomy.

DETAILED DESCRIPTION:
The study will be in 3 parts:

First one will be to address the key question of the lower limb frontal alignment based on both three-dimensional measurements of low-dose bi-planar X-rays and foot morphology assessment. Indeed, a major issue in the management of lower limb disorders is the ability to correctly assess abnormal development and decide on the most adapted treatment option. In particular, the link between lower limb disorders and foot morphology remain unclear. Recently, quantitative 3D measurement of the lower limb in children has been successfully assessed using low-dose biplanar X-rays. The population studied will be 133 patients, aged 6 to 16 years old, for whom a lower limb standing X-ray is required for a medical reason not interfering with torsional or longitudinal axis of the limb (such as, for example, patients consulting for non-specific lower limb pain). All patients will have low-dose biplanar X-rays using the EOS® system (EOS® Imaging, France). From the EOS® bi-planar images, a 3D patient-specific parametric model of the lower limbs will be obtained. The clinical indices (i.e. mechanical femoral (MFA) and mechanical tibial (MTA) angles, Hip Knee Shaft angle (HKS) and femoro tibial angle (FTA)) will then be automatically computed. For each clinical parameter, the mean value and standard deviation will be calculated, depending on the age group, gender, and on foot morphology

Second part is to assess the reproducibility of the 3dimensional reconstructions whether they are made by a radiology technician, or by a so-called expert through collecting datas from 3 centers of pediatric surgery where EOS Imaging system is daily used to get spine or lower limb X-Rays. The investigators will include 20 children, divided as follow: six typically developing ones (control X-Rays or lower limb standing X-ray required for a medical reason not interfering with torsional or longitudinal axis of the limb), 6 non-typically developing (by example children who underwent a lower limb fracture), 6 cerebral palsy ones, and 2 children with extreme lower limb deformities. Reconstructions will be done twice in each center: once by a qualified operator, senior orthopedic surgeon, who followed a practical course, and once by a radiology technician, also used to the software.

First step will be to calculate the reproducibility for all parameters, depending on each subgroup of patient. Then, for each parameter, outliers' values will be analyzed and explained. They will be then suppressed from the datas to re-calculate the reproducibility. Finally, reproducibility of the obtained parameters will be compared to the one published in literature

Last part will be to work on the recently developed weight-bearing foot 3D reconstruction method for clinical use using the Parametric Personalized Modelling approach (PPM). This will allow having a better understanding and evaluation of foot's anatomy and patho-anatomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 6 and 18 years, feminine and male. -Preliminary clinical examination - Statigramme by the system EOS ® (pond shin thighbone foot) prescribes within the framework of a surveillance of any pathology not interfering with the data to be studied
* Patients capable of standing without moving and without help the time of the acquisition EOS ®, approximately 30 seconds.
* Consent of the patient and the legal representative
* Membership in a national insurance scheme

Exclusion Criteria:

* Child before 6 years or after 18 years
* Incapacitated to stand(to hold water) without support(medium) and without moving during 30 seconds (time(weather) of acquisition Of the image)
* History of pathology or surgical gesture(movement) on lower limbs which can modify Frontal bone or the twistings of lower limbs morphotype.
* Refusal of the legal representative or the patient.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 83 (Actual)
Dates: Start 2014-05-25 (Actual); Primary Completion 2016-05-20 (Actual); Study Completion 2016-05-20 (Actual)

PRIMARY OUTCOMES:
3D reconstruction of the angle of the lower limb | At baseline during the visit of inclusion
  The modelling in 3 D lower limbs will be made from the following measures on the acquisitions of lower limbs:
  *In the frontal plan (face) mechanical angles:
  Angle LPFA: side femoral proximal angle: 90 ° (85-95 °) mLDFA angle: side mechanical femoral distal angle 87 ° (85-90 °) angle MPTA: medial proximal tibial angle: 87 ° (85-90 °) angle LDTA: side distal tibial angle: 89 ° (86-92 °) anatomical angles:
  Angle HKA: center of the femoral head centers of the knee center of the ankle: 176-180 ° angle MPFA: femoral medial proximal angle: 84 ° (80-89 °) aLDFA angle: side anatomical femoral distal angle: 81 ° (79-83 °) angle MPTA: medial proximal tibial angle: 87 ° (85-90 °) angle LDTA: side distal tibial angle: 89 ° (86-92 °) *In the saggital plan (profile): Angle PDFA: femoral posterior distal angle: 83 ° (79-87 °) angle PPTA: posterior proximal tibial angle: 81 ° (77-84 °) angle ADTA: anterior distal tibial angle: 80 ° (78-82 °)
  *In the horizontal plan: Femoral twisting 7-24 °

SECONDARY OUTCOMES:
3D reconstruction of the angle of lower limbs according to age group | At baseline during the visit of inclusion
  To study the model in 3D of lower limbs according to age group (6-9 years; 10-12 years; 13-15 years; 16-18 years)
  The modelling will be made from the following measures :
  *In the frontal plan mechanical angles:
  Angle LPFA: side femoral proximal angle: 90 ° (85-95 °), side mechanical femoral distal angle 87 ° (85-90 °), angle medial proximal tibial angle: 87 ° (85-90 °), side distal tibial angle: 89 ° (86-92 °) anatomical angles:
  Center of the femoral head centers of the knee center of the ankle: 176-180 ° angle femoral medial proximal angle: 84 ° (80-89 °), side anatomical femoral distal angle: 81 ° (79-83 °) angle medial proximal tibial angle: 87 ° (85-90 °), side distal tibial angle: 89 ° (86-92 °) *In the saggital plan (profile): Angle femoral posterior distal angle: 83 ° (79-87 °) angle posterior proximal tibial angle: 81 ° (77-84 °) angle anterior distal tibial angle: 80 ° (78-82 °)
  *In the horizontal plan: Femoral twisting 7-24 °
Valuable elaboration in 3 dimensions of the angle to characterize the various groups of feet | At baseline during the visit of inclusion
  Valuable elaboration in 3 dimensions(size) to characterize the various groups of feet by measuring on the reconstructions obtained from the following already known angles:
  Picture dorso plantar:
  talocalcaneal difference: longitudinal axis bank and calcaneus 15-25 °. Talus Angle - 1st metatarsal: 0 10 °. Angle calcaneus - 5th metatarsal: 0 °. talo navicular cover Angle : median longitudinal axis of the bank and perpendicular in the frontal axis of the naviculaire.
  Cuneo angle-M1: perpendicular in the edge medial of the medial cuneiform and space cm M1: 10-20 °.
  Report column medial (calca médial + M1) / side column (calca side + M5): Men: 26, Women: 34 (between 5 and 17 years).

CONTACTS AND LOCATIONS:
Overall Officials: Virginie RAMPAL, MD, Principal Investigator — Fondation Lenval
Locations (2):
- France (2):
  - Fondation Lenval, Nice
  - Hôpital Necker enfants Malades, Paris